CLINICAL TRIAL: NCT02928523
Title: PreventiOn of DYSbioSis Complications With Autologous Fecal Microbiota Transplantation in acutE myEloid Leukemia Patients Undergoing Intensive Treatment: A Feasibility and Safety Study ODYSSEE STUDY
Brief Title: PreventiOn of DYSbioSis Complications With Autologous FMT in AML Patients
Acronym: ODYSSEE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPOH02
Record Dates: First submitted 2016-05-26; First posted 2016-10-10 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Autologous Fecal Microbiota Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Fecal Microbiota Transplantation (Experimental): Patients will receive autologous fecal microbiota transplantation (MaaT011- 150 mL rectal enema) - 2 administrations 24 hours apart.
  Interventions: Drug: Autologous Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Autologous Fecal Microbiota Transplantation
  Other Names: MaaT011

SUMMARY:
The investigators propose to use autologous fecal microbiota transplantation (AFMT) to acute myeloid leukemia (AML) patients treated with intensive chemotherapy and antibiotics in order to restore the balance of their intestinal microbiome and thereby eradicate treatment-induced multidrug resistant bacteria (MDRB), infection-related complications, as well as sequelae to the gastrointestinal tract. Therefore, the investigators propose to perform a single-arm multicentre prospective fecal microbiota transplantation (FMT) trial in AML patients receiving intensive chemotherapy, and who are usually heavily treated with broad-spectrum antibiotics during aplasia that generate a profound status of dysbiosis. For this purpose, at the time of admission and AML diagnosis, patients will be requested to donate stools that will be comprehensively screened, and if deemed appropriate according to protocol criteria, conditioned and stored frozen until future processing and transplantation after aplasia completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤ 75 years old with de novo diagnosis of AML or high-risk myelodysplastic syndrom for whom intensive induction chemotherapy is anticipated within 10 days after admission
* Patients willing to donate stool samples and to follow protocol recommendations
* Signature of informed and written consent

Exclusion Criteria:

* Acute promyelocytic leukemia (AML-M3)
* Known allergy or intolerance to trehalose or maltodextrin
* Pregnancy: positive urinary or blood test in female of childbearing potential
* Severe disease with a life expectancy < 3 months
* Other ongoing interventional protocol that might interfere with the study
* Non eligibility for collection of autologous stools upon admission:

  * Patients refusing to consent
  * Antibiotherapy at the time of study inclusion ≥ 4 days
  * Concomitant or previous diagnosis of a significant inflammatory bowel disease (UC, CD) or other progressive digestive disease requesting treatment or further medical exploration
  * Presence of severe colitis of any etiology at the time of admission or severe digestive disorders (acute or chronic diarrhea) within 3 months preceding inclusion
  * Patient getting a recent colonoscopy (within 3 months preceding inclusion)
* Detection of MDRB, pathogenic bacteria, parasites, norovirus and/or rotavirus during screening of autologous stool collected at baseline
* Non eligibility for inoculum transplantation: persistent mucositis, colitis, or haemorrhoids, presence of blood in more than 50% of patient's faeces the week preceding the transplantation
* Non feasibility of inoculum procedure: patient refusal; technical or biological mismatch of the inoculum
* Absence of effective contraceptive method for female of childbearing potential
* Lactation
* Inability to give an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of AFMT efficacy in dysbiosis correction by measure of microbiota diversity | 40 days
  Comparison of Alpha and Beta diversity indexes at baseline, after chemotherapy and after AFMT will be performed
Evaluation of AFMT efficacy in MDRB eradication based on bacterial culture | 40 days
  MDRB carriage and resistome will be compared at baseline, after chemotherapy and after AFMT

SECONDARY OUTCOMES:
Definition of a dysbiosis biosignature using combination of biological parameters | 40 days
  Microbiota sequencing results will be correlated with immune parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, MD, PhD, Study Chair — APHP
Locations (4):
- France (4):
  - IPC, Marseille
  - CHU Nantes, Nantes
  - Hopital Saint Antoine, Paris
  - HCL Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malard F, Vekhoff A, Lapusan S, Isnard F, D'incan-Corda E, Rey J, Saillard C, Thomas X, Ducastelle-Lepretre S, Paubelle E, Larcher MV, Rocher C, Recher C, Tavitian S, Bertoli S, Michallet AS, Gilis L, Peterlin P, Chevallier P, Nguyen S, Plantamura E, Boucinha L, Gasc C, Michallet M, Dore J, Legrand O, Mohty M. Gut microbiota diversity after autologous fecal microbiota transfer in acute myeloid leukemia patients. Nat Commun. 2021 May 25;12(1):3084. doi: 10.1038/s41467-021-23376-6. PMID 34035290